CLINICAL TRIAL: NCT02507609
Title: The Effect of Deep Neuromuscular Block on Cytokines Release and Postoperative Delirium of Elderly Patients Undergoing Total Hip Arthroplasty
Brief Title: Deep Neuromuscular Block on Cytokines Release and Postoperative Delirium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Konkuk University Medical Center (Other)
Responsible Party: Principal Investigator, Seong-Hyop Kim, Associate Professor, Konkuk University Medical Center
Allocation: Randomized | Model: Factorial | Masking: Quadruple | Purpose: Treatment
Other Study IDs: KUH1160087
Record Dates: First submitted 2015-07-21; First posted 2015-07-24 (Estimated); Last update posted 2018-06-20 (Actual); Status verified 2018-06

CONDITIONS: Hip Fractures
MeSH Terms: conditions — Hip Fractures | interventions — Rocuronium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- M group (Active Comparator): moderate neuromuscular blockade group by intermittent injection of rocuronium bromide
  Interventions: Other: Moderate neuromuscular blockade
- D group (Active Comparator): deep neuromuscular blockade group by continuous infusion of rocuronium bromide
  Interventions: Other: Deep neuromuscular blockade

INTERVENTIONS:
Other: Moderate neuromuscular blockade — TOF count is maintained to 1 to 2 by intermittent intravenous injection of rocuronium bromide 5 mg during operation
  Other Names: Esmeron
  Arms: M group
Other: Deep neuromuscular blockade — PTC is maintained to 1 to 2 degree by continuous infusion of rocuronium bromide intravenous route
  Other Names: Esmeron
  Arms: D group

SUMMARY:
The purpose of the study is to determine the relationship between the degree of neuromuscular block, the release of cytokines and clinical outcomes in elderly patients undergoing orthopedic surgery. Investigators hypothesize that deep neuromuscular blockade decreases the release of cytokine and the incidence of postoperative delirium in elderly patients undergoing orthopedic surgery, compared with moderate neuromuscular blockade.

DETAILED DESCRIPTION:
* Study design

  - This is a prospective, randomized, single blinded study.
* Measurement values

  * Neuromuscular monitoring by post-tetanic count (PTC) during operation
  * Regional cerebral oxygen saturation monitoring
  * Mean systemic blood pressure (MBP), heart rate (HR)
  * Cardiac index (CI), using non-invasive cardiac output monitor
  * IL-1ß, IL-6, TNF-α, IL-10 and CRP
  * Arterial blood gas analysis (ABGA)
  * Laboratory values [Hemoglobin, Hematocrit, serum albumin, creatinine, CPK, LDH]
  * Postoperative pain, using visual analogue scale (VAS)
  * Postoperative nausea and vomiting (PONV)
  * Total infused amounts of drugs
  * Total anesthesia duration, intubation duration and operation duration
  * Intubation duration, operation duration
  * Incidence of postoperative intensive care unit (ICU) admission
  * Total ICU staying duration, if patients admit to ICU
  * Preoperative and postoperative left ventricular ejection fraction change
  * Incidence of hypotension (mean blood pressure lesser than 60 mmHg)
  * Incidence of postoperative delirium using confusion assessment method (CAM) intensive care unit (ICU)
  * Total amount of blood products transfusion (paced red blood cells, fresh frozen plasma, platelet concentration, cryoprecipitate)
  * Total amount of crystalloids and colloids infusion
  * Total amount urine output

ELIGIBILITY:
Inclusion Criteria:

* All adult (more than 50 years old) patients scheduled for total hip arthroplasty and total knee arthroplasty who have signed the written informed consent.

Exclusion Criteria:

* Inability to give informed consent
* Preexisting cognitive dysfunction or delirium
* Known allergy to rocuronium sugammadex
* Underlying liver dysfunction (AST and ALT more than 100 IU/l)
* Underlying kidney dysfunction (Serum Creatinine more than 1.5 mg/dl)
* Underlying neuromuscular disease
* Patients taking any medication with potential interference with neuromuscular transmission

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 82 (Actual)
Dates: Start 2015-09-08 (Actual); Primary Completion 2018-04-26 (Actual); Study Completion 2018-04-26 (Actual)

PRIMARY OUTCOMES:
Interleukin 6 | postoperative 4 hours

SECONDARY OUTCOMES:
postoperative delirium | up to postoperative day 7
  The incidence of postoperative delirium will be assessed by using confusion assessment method (CAM)

CONTACTS AND LOCATIONS:
Overall Officials: Seong-Hyop Kim, M.D., Principal Investigator — Konkuk University Medical Center
Locations (1):
- Konkuk University Medical Center, Seoul, South Korea

REFERENCES:
- [Derived] Oh CS, Lim HY, Jeon HJ, Kim TH, Park HJ, Piao L, Kim SH. Effect of deep neuromuscular blockade on serum cytokines and postoperative delirium in elderly patients undergoing total hip replacement: A prospective single-blind randomised controlled trial. Eur J Anaesthesiol. 2021 Mar 1;38(Suppl 1):S58-S66. doi: 10.1097/EJA.0000000000001414. PMID 33399376